CLINICAL TRIAL: NCT03002428
Title: A Randomized Study Comparing the Effects of PF708 and Forteo in Patients With Osteoporosis
Brief Title: A Comparison of PF708 and Forteo in Osteoporosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfenex, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF708-301
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (PF708) (Experimental): PF708 20 mcg once-daily subcutaneous injection for 24 weeks
  Interventions: Drug: Teriparatide (PF708)
- Teriparatide (Forteo) (Active Comparator): Forteo 20 mcg once-daily subcutaneous injection for 24 weeks
  Interventions: Drug: Teriparatide (Forteo)

INTERVENTIONS:
Drug: Teriparatide (PF708) — Subcutaneous injection
  Arms: Teriparatide (PF708)
Drug: Teriparatide (Forteo) — Subcutaneous injection
  Arms: Teriparatide (Forteo)

SUMMARY:
The purpose of this study is to compare the effects of two teriparatide products, PF708 and Forteo, in patients with osteoporosis.

DETAILED DESCRIPTION:
This is a randomized, multi-center study conducted in the United States. Men and women with osteoporosis will be enrolled in a parallel-group, open-label study design to compare the effects of PF708 and Forteo after 24 weeks of treatment. Half of the subjects will be randomized to receive PF708, and the other half will be randomized to receive Forteo.

ELIGIBILITY:
Inclusion Criteria:

* If female, ≥5 years postmenopausal at the time of screening, with a DXA-derived BMD value at least 1 standard deviation (SD) below the average of young, healthy women
* If male, has a DXA-derived BMD value at least 2 SD below the average of young, healthy men
* Able to use the pen injection device correctly
* Able to understand and sign the written Informed Consent Form (ICF)

Exclusion Criteria:

* Treatment with oral bisphosphonates (once daily or once weekly) within 6 months of screening
* Any current or prior human PTH-derived products (e.g., Forteo, Teribone, Natpara), including for investigational purposes
* Immobility due to severe or chronically disabling conditions (e.g., stroke, Parkinson's disease, multiple sclerosis)
* History of metabolic bone diseases other than osteoporosis
* History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured)
* History of Paget's disease of bone
* History of prior external beam or implant radiation therapy involving the skeleton
* Active urolithiasis or primary hyperparathyroidism

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Blood levels of anti-drug antibody (ADA) against teriparatide | 24 weeks

SECONDARY OUTCOMES:
Mean percentage change in lumbar-spine bone mineral density (BMD) | 24 weeks
Median percentage change in serum N-terminal propeptide of type 1 procollagen (P1NP) | 24 weeks
Median percentage change in serum crosslinked C-terminal telopeptide of type 1 collagen (CTX) | 24 weeks
Plasma maximum concentration (Cmax) of teriparatide | 4 hours
Plasma area-under-the-curve (AUC) of teriparatide | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hubert C Chen, MD, Study Director — Pfenex, Inc
Locations (25):
- United States (25):
  - Radiant Research, Birmingham, Alabama
  - The Orthopaedic Group, Mobile, Alabama
  - Radiant Research, Chandler, Arizona
  - Radiant Research, Mesa, Arizona
  - SunValley Arthritis Center, Peoria, Arizona
  - Radiant Research, Phoenix, Arizona
  - Radiant Research, Colorado Springs, Colorado
  - OB-GYN Associates of Mid-Florida, Leesburg, Florida
  - Atlanta Research Center, Atlanta, Georgia
  - Radiant Research, Chicago, Illinois
  - Radiant Research, Bridgeton, Missouri
  - Radiant Research, Papillion, Nebraska
  - Radiant Research, Henderson, Nevada
  - Radiant Research, Las Vegas, Nevada
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Lillestol Research, Fargo, North Dakota
  - Radiant Research, Akron, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Pennsylvania Regional Center for Arthritis & Osteoporosis Research, Wyomissing, Pennsylvania
  - Radiant Research, Dallas, Texas
  - Radiant Research, Plano, Texas
  - Radiant Research, San Antonio, Texas
  - Spectrum Medical, Danville, Virginia
  - Radiant Research, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No